CLINICAL TRIAL: NCT04338724
Title: A Phase I, Open-Label, Dose-Escalation Study of the Anti-CTLA-4 Monoclonal Antibody CS1002 in Subjects With Advanced Solid Tumors
Brief Title: A Phase I Study of CS1002 in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CStone Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CS1002-102
Record Dates: First submitted 2020-03-31; First posted 2020-04-08 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CS1002 (Experimental)
  Interventions: Drug: CS1002

INTERVENTIONS:
Drug: CS1002 — The dose levels will be escalated following a modified 3+3 dose escalation scheme.

SUMMARY:
This is an open label, dose escalation phase I study to evaluate the clinical safety, tolerability in subjects with advanced solid tumors, and to establish the Maximum Tolerated Dose (MTD#, if any). This study is composed of two dose level: 1 and 3 mg/kg.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent for the study.
2. Being ≥18 years of age on the day of signing informed consent.
3. Subjects must have a histologically or cytologically confirmed advanced or metastatic solid tumor(s) for which no effective standard therapy is available or tolerable.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
5. Subjects with evaluable but non-measurable lesion are allowed to participate in the study.
6. Life expectancy ≥12 weeks.
7. Subject must have adequate organ function as indicated by laboratory values
8. Fertile men and women of childbearing potential must agree to use an effective method of birth control from providing signed consent and for 180 days after last investigational product administration. Women of childbearing potential include pre-menopausal women and women within the first 2 years of the onset of menopause. Women of childbearing potential must have a negative pregnancy test ≤ 7 days prior to the first dose of investigational product.

Exclusion Criteria:

The subject must be excluded from participating in the study if the subject:

1. Known brain metastasis, primary central nervous system (CNS) or another CNS metastasis that is either symptomatic or untreated. Central nervous system metastases that have been treated by complete resection and/or radiotherapy demonstrating stability or improvement are not an exclusion criterion provided they are stable as shown by imaging for at least 4 weeks before Screening without evidence of cerebral edema and no requirements for corticosteroids or anticonvulsants.
2. Subjects with active autoimmune diseases or a history of autoimmune diseases should be excluded; these include but are not limited to subjects with a history of immune-related neurologic disease, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barre syndrome, myasthenia gravis, systemic lupus erythematosus, connective tissue diseases, scleroderma, inflammatory bowel disease including Crohn's disease and ulcerative colitis, hepatitis, toxic epidermal necrolysis, Stevens-Johnson syndrome, or antiphospholipid syndrome.
3. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy (eg, >10 mg daily prednisone equivalents) or any other form of immunosuppressive therapy within 14 days prior to the Cycle 1 Day 1. The use of physiologic doses of corticosteroids may be approved after consultation with the Sponsor.
4. Has received prior therapy with an anti-CTLA-4 agent.
5. Has had prior chemotherapy, targeted therapy, or any other agents used as a systemic treatment for cancer, within 21 days of Cycle 1 Day 1
6. Known history of human immunodeficiency virus (HIV) infection.
7. Active tuberculosis infection.
8. Subjects with a known history of alcoholism or drugs abuse.
9. Subjects with the major cardiovascular condition (eg, congestive heart failure, unstable angina pectoris, atrial fibrillation, arrhythmia.): subjects who had experienced such conditions such as acute myocardial infarction, unstable angina pectoris, apoplexia, or transient ischemic attack within 6 months prior to Cycle 1 Day 1; subjects with congestive heart failure of New York Heart Association Grade ≥2.
10. Concurrent condition that in the investigator's opinion would jeopardize compliance with the protocol.
11. Unwillingness or inability to follow the procedures outlined in the protocol.
12. Women with pregnancy or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-12-27 (Actual); Primary Completion 2020-09-21 (Actual); Study Completion 2020-09-21 (Actual)

PRIMARY OUTCOMES:
safety and tolerability | From the day of first dose to 21 days after last dose
  Number of participants with adverse events
area under the curve | From the time of infusion to 21 days after first dose and forth dose
  (AUC)0-21d
maximum observed serum concentration (Cmax) | From the time of infusion to 21 days after first dose and forth dose

CONTACTS AND LOCATIONS:
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China